CLINICAL TRIAL: NCT07318402
Title: Operator Radiation Exposure During Image-Guided Robotic-Assisted Bronchoscopy: A Multicenter Prospective Cohort Study
Status: Recruiting | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 25-350
Record Dates: First submitted 2025-12-23; First posted 2026-01-06 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Operator Radiation Exposure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Operator Radiation: During Image-Guided Robotic-Assisted Bronchoscopy

SUMMARY:
This is a multicenter, single-arm, prospective, observational study designed to evaluate bronchoscopist radiation exposure during standard-of-care image-guided robotic-assisted bronchoscopy (RAB) for sampling of a single pulmonary parenchymal lesion.

ELIGIBILITY:
Inclusion Criteria:

* Operator performing image-guided RAB on adult patients (age ≥18 years old)
* A single participating operator per study site
* Image-guided RAB procedure is planned for standard of care diagnostic sampling of a single parenchymal lung lesion at participating sites

Exclusion Criteria:

* Operator refusal to participate
* Image-guided RAB procedure performed on:

  * Patients age <18 years old
  * Pregnant women
  * Patients undergoing standard of care robotic assisted bronchoscopy with plan to sample >1 pulmonary parenchymal lesion
  * Patients undergoing standard of care robotic assisted bronchoscopy for lesion localization (injection of dye/marker or fiducial marker deployment)
  * Patients undergoing standard of care robotic assisted bronchoscopy for a therapeutic intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Operator performing standard of care image-guided robotic-assisted bronchoscopy for the sampling of a single pulmonary parenchymal lesion
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2025-12-23 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
total operator radiation exposure dose | 1 year
  as captured by a radiation dosimetry badge over 50 consecutive procedures. All study procedures in which image-guided RAB was performed for the sampling of a single parenchymal lung lesion will be evaluable for the primary endpoint.

CONTACTS AND LOCATIONS:
Overall Officials: Or Kalchiem-Dekel, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan Kettering Cancer Center (All Protocol Activites), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — https://www.mskcc.org